CLINICAL TRIAL: NCT04183270
Title: BELgian ANtiCOagulation Survey for NVAF Patients
Brief Title: Survey on Belgian Patients Suffering From Irregular Heartbeat and Starting Treatment With a Drug to Prevent Blood Clots in Blood Vessels and the Heart. This Study is Also Called BELANCOS.
Acronym: BELANCOS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21153
Record Dates: First submitted 2019-11-21; First posted 2019-12-03 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Non-valvular atrial fibrillation (NVAF) patients who will start treatment with a non-VKA oral anticoagulants (NOAC).
  Interventions: Other: Questionnaires
- Physicians: Treating physicians for NVAF patients.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — The survey will focus on non-valvular atrial fibrillation patients, who will start treatment with a NOAC, and their treating physician.

SUMMARY:
In this study researchers want to learn more about the patient's and treating doctor's concerns about possible bleedings during treatment with drugs preventing blood clots in blood vessels and the heart - so called blood thinner. The study also wants to find out more about the patient's knowledge on the importance, risks and benefits of treatment with this drug group.

Patients with irregular heartbeat not caused by valvular heart disease who will start treatment with a blood thinner will be asked by their treating cardiologist to complete a questionnaire related to their knowledge and fear of possible bleedings or stroke (blockage or rupture of a blood vessel to the brain) due to the intake of a blood thinner. The treating doctor will complete a similar questionnaire. The study plans to involve 15 cardiologists and 300 patients in Belgium.

ELIGIBILITY:
Inclusion criteria:

* Male or female adult patients diagnosed with NVAF.
* NOAC treatment-naive patients who will start a NOAC treatment.

Exclusion criteria:

* Previous stroke or thrombosis
* Previous severe bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population of this study would be approximately 15 cardiologists (hospital or office-based) and 300 NOAC treatment-naïve patients diagnosed with NVAF who will start treatment with a NOAC for this indication.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Age categories of patients | 1 day
  Collected via the questionnaire.
Gender (Female or male) of patients | 1 day
  Collected via the questionnaire.
Patients' level of agreement with various statements of using NOACs in general | 1 day
  By using a 5-point Likert scale (completely disagree, more likely to disagree, no opinion, more likely to agree, completely agree)
Level of patients fear of having a bleeding on a scale from 0 - 10 | 1 day
Level of patients fear of having a stroke or thrombosis on a scale from 0 - 10 | 1 day
Age categories of physicians | 1 day
  Collected via the questionnaire.
Gender (Female or male) of physicians | 1 day
  Collected via the questionnaire.
Physicans' level of agreement with various statement of using NOACs in general | 1 day
  By using a 5-point Likert scale (completely disagree, more likely to disagree, no opinion, more likely to agree, completely agree)
Level of patients fear of having a bleeding assessed by physicans on a scale from 0 - 10 | 1 day
Level of patients fear of having a stroke or thrombosis assessed by physicians on a scale from 0 - 10 | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Belgium

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.